CLINICAL TRIAL: NCT04732884
Title: A Prospective Randomized Controlled Monocentric Trial Evaluating the Effect of Biofeedback on Osseous Union Using Pedobarography After Mid- and Hindfoot Arthrodesis
Brief Title: Evaluation of the Effect of Biofeedback on Osseous Union Using Pedobarography After Mid- and Hindfoot Arthrodesis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was suspended for technical reasons
Sponsor: Prof. Dr. med. Arno Frigg (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Arno Frigg, Prof. Dr. med., Klinik Hirslanden, Zurich
Organization: Klinik Hirslanden, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BioPed
Record Dates: First submitted 2021-01-09; First posted 2021-02-01 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Complication of Surgical or Medical Care
Keywords: mid- and hindfoot surgical arthrodesis; osseous non-union
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Radiologists assessing the primary outcome osseous non-union will be blind to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight sensor with biofeedback (Experimental): Activation of the feedback function of the weight-bearing sensor as mean to possibly enhance compliance to weight-bearing instructions postoperative.
  Interventions: Device: Smartsens, Gelenic AG; with biofeedback
- Weight sensor without biofeedback (Experimental): Standard patient education considering postoperative weight-bearing parameters and measurement of actual weight-bearing with the sensor.
  Interventions: Device: Smartsens, Gelenic AG; without biofeedback

INTERVENTIONS:
Device: Smartsens, Gelenic AG; with biofeedback — The Smartsens is a CE certified 4-cell load sensor integrated in an insole that can be placed in any orthosis or cast. A threshold (10-50kg) can be defined at which - if higher loads are measured - an audio signal warns the patient of overloading (biofeedback). The device additionally registers loads from 0-100kg continuously.
  Other Names: Weight sensor with biofeedback
  Arms: Weight sensor with biofeedback
Device: Smartsens, Gelenic AG; without biofeedback — Patients will not be warned by an audio signal in case of overloading. The device registers loads from 0-100kg continuously.
  Other Names: Weight sensor without biofeedback
  Arms: Weight sensor without biofeedback

SUMMARY:
The current study aims at evaluating the effect of biofeedback of correct partial weight bearing on the rate of osseous non-union compared to conventional patient instruction without biofeedback.

DETAILED DESCRIPTION:
Post-traumatic situations or instabilities of other aetiology at the level of the foot can lead to painful degenerative arthritis that necessitates surgical arthrodesis for pain relief. Surgical arthrodesis in this region though is associated with a high risk of osseous non-union (depending on the exact location up to 40%) despite standardized preparation and fixation techniques. The development of osseous non-union is associated with certain patient characteristics like active smoking, nutrition etc. Compliance to partial weight-bearing during the early postoperative phase is another contributing factor.

The current study aims at evaluating the effect of biofeedback of correct partial weight bearing on the rate of osseous non-union compared to conventional patient instruction without biofeedback.

All patients will postoperatively be provided with a lower- leg unloading orthosis furnished with a weight sensor that will - according to randomization - give feedback if a predefined weight threshold has been crossed or just measure weight-bearing without feedback.

ELIGIBILITY:
Inclusion Criteria:

* Indication for hind- or midfoot arthrodesis
* Informed Consent
* Body weight < 90kg (according to Smartsens manufacturers recommendations)

Exclusion Criteria:

* Physical or mental inability to follow weight-bearing recommendations (e.g. dementia, neurologic disease, upper extremity pathology)
* Participation in a potentially interfering interventional trial during the last 30 day or before wash-out of any trial medication (e.g. steroids, medications affecting bone metabolism etc.)
* Previous infection at the intended surgical site
* Body weight > 90kg
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the influence of weight bearing an resting time on the development of osseous non-union after surgical arthrodesis at the level of the mid- and hindfoot. | 3 months
  The primary outcome is an analysis of the rate of non-unions after mid- and hindfoot arthrodesis comparing a sensor the two patient arms with activated vs non-activated biofeedback.
  The rate of osseous non-unions defined as CT-morphologic union <30% of the joint surface at 3 months in relation to the provision of biofeedback.

SECONDARY OUTCOMES:
Compliance i.e. adherence to weight bearing recommendations (≤ 15kg charge) with and without biofeedback. | 6 weeks
  All patients will be asked to wear the orthosis with integrated sensor all day long including resting times. They are furthermore instructed to follow partial weight-bearing with 15kg (for 6 weeks).
  The device will record load and quantity of steps over time. In the first group, a biofeedback in form of an audio-signal will warn the patient if treatment recommendations like partial weight bearing are not followed. The control intervention will be pure instruction followed by measurements. Control patients will not receive biofeedback upon transgression of recommendations.
Compliance i.e. adherence to resting time recommendations (≥ 80% of time) with and without biofeedback. | 6 weeks
  All patients will be asked to wear the orthosis with integrated sensor all day long including resting times. They are furthermore instructed to reduce their activity with 80% resting time.
  The device will record load and quantity of steps over time. In the first group, a biofeedback in form of an audio-signal will warn the patient if treatment recommendations like resting times are not followed. The control intervention will be pure instruction followed by measurements of load and quantity of steps. Control patients will not receive biofeedback upon transgression of recommendations.
Consumption of analgesic medication after surgery | 12 months
  Consumption of analgesic medication following WHO grading. Data will be collected at any scheduled (2 and 6 weeks, 3 and 12 months) or unscheduled follow-up visits.
Patient's quality of life after surgery | 12 months
  Quality of life will be analysed by using EuroQuality of Life Five Dimensions (EQ5D-5L) questionnaire at baseline and after 3 months and 12 months.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Patient's satisfaction | 12 months
  Patient satisfaction will be documented after 2 weeks, 6 weeks, 3 months and 12 months by using net promotor score (NPS).
  NPS is the percentage of customers rating their likelihood to recommend the "service" to a friend or colleague as 9 or 10 ("promoters") minus the percentage rating this at 6 or below ("detractors") on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- FussZentrumHirslanen, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No